CLINICAL TRIAL: NCT05302778
Title: Observational Study Evaluating the Role of Eribulin as a Second-line Treatment in Triple-negative Advanced Breast Cancer
Brief Title: Eribulin as a Second-line Treatment in Triple-negative Advanced Breast Cancer
Acronym: HERMIONE-10
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Collaborators: EISAI s.r.l. (Unknown)
Responsible Party: Sponsor
Other Study IDs: HERMIONE-10
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Triple Negative Breast Cancer
Keywords: breast cancer; triple negative; second line; eribulin; real world
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter, retrospective and prospective, cohort, observational study evaluating the clinical efficacy and tolerability of Eribulin as second-line treatment in accordance with the indications authorized by AIFA in patients with triple negative advanced breast cancer in a real world setting.

DETAILED DESCRIPTION:
The study, multicenter, retrospective and prospective, cohort, observational, describes the modalities of treatment with Eribulin as a second line therapy for triple negative breast cancer and "clinical outcomes" in a population real-world, evaluating any differences with the results obtained in clinical trials. Therapeutic sequences will also be evaluated with the aim of providing a photograph of the choices made in clinical practice in this historical moment characterized by rapid evolution of new molecules available to clinicians.

A total of at least 200 patients with triple negative advanced breast cancer treated with Eribulin as second line will be enrolled in the retrospective or prospective cohort. Enrollment period will last 2 years.

Pseudoanonymized data will be collected in a electroctronic database (RedCap Cloud); here the list of the main variables collected:

* Patient Registration
* Demography
* Pregnancy test
* Past history and habits of the patient
* Previous antineoplastic therapy
* Anamnesis close to entering the study
* Vital signs and ECOG performance status (WHO)
* Blood chemistry tests
* RECIST 1.1 Baseline and re-evaluations
* 12 Lead ECG evaluation
* Eribulin cycles
* Adverse events
* Previous and concomitant medications
* End of study

The retrospective analysis of the choices made in clinical practice and the benefits obtained from the second therapeutic lines could provide important data to favor the definition of prospective randomized studies, and guide the clinician towards a better therapeutic path.

ELIGIBILITY:
Inclusion Criteria:

* Performance status according to ECOG equal to 0-2
* Locally advanced or triple negative metastatic breast cancer (HR- and HER2-) confirmed histologically
* Progressing after first-line chemotherapy for advanced disease
* Previous anthracyclines and taxanes therapy (in an adjuvant, neoadjuvant or metastatic), unless the patient is ineligible to receive such treatments
* Treatment with Eribulin mesylate since 2017, in accordance with AIFA indications
* Adequate haematological, renal and hepatic function, as per clinical practice
* Written informed consent

Exclusion Criteria:

* Breast cancer HER2 + or HR +
* Treatment with Eribulin in the context of clinical studies
* Patients unsuitable for treatment with Eribulin
* Diagnosis of other malignancies in the two years prior to enrollment, with one exception of adequately treated localized basal cell or squamous cell carcinomas of the skin o cervical carcinomas undergoing curative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic triple negative breast cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Entire study duration, approximately 3 years
  PFS defined as time from the beginning of treatment to disease progression or death

SECONDARY OUTCOMES:
Time to progression (TTP) | Entire study duration, approximately 3 years
  TTP defined as the time from the beginning of treatment to disease progression or death
Overall Response Rate (ORR) | Entire study duration, approximately 3 years
  OOR defined as the percentage of patients who achieved a partial response (PR) or a complete response (CR) as best response according to RECIST 1.1
Disease Control Rate (DCR) | Entire study duration, approximately 3 years
  DCR defined as the percentage of patients who achieved a partial response (PR), a complete response (CR) or a stable disease (SD) as best response according to RECIST 1.1 criteria, according to the site of metastatic disease (bone disease vs visceral disease with or without bone involvement).
Site of progression | Entire study duration, approximately 3 years
  Description of sites of progression in patients with first bone relapse
Duration of response and disease control | Entire study duration, approximately 3 years
  Duration of response and disease control
Survival after progression | Entire study duration, approximately 3 years
  Survival after progression
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Entire study duration, approximately 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - ASST Monza, Monza
  - Oncologia Medica Policlinico Universitario Palermo, Palermo
  - OSPEDALE LA MADDALENA, Palermo, Palermo